CLINICAL TRIAL: NCT00565058
Title: A Phase II Simon Two-stage Multicenter Study and Pilot Pharmacodynamic Investigation of GTI 2040 in Combination With High Dose Cytarabine (HiDAC) in Refractory and Relapsed Acute Myeloid Leukemia (AML)
Brief Title: Combination of GTI-2040 and Cytarabine in the Treatment of Refractory and Relapsed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aptose Biosciences Inc. (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2040AML201
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — GTI2040

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilot (Experimental): Pilot PD Study (Delayed GTI-2040) Group: In the Pilot PD Study Group, addition of GTI-2040 is delayed until 24 hours after initiation of HiDAC.
  Interventions: Biological: GTI-2040
- Phase II arm (Experimental): Phase II PD Study (Early GTI-2040) Group: In the Phase II PD Study Group, GTI-2040 is given 24 hours prior to addition of HiDAC.
  Interventions: Biological: GTI-2040

INTERVENTIONS:
Biological: GTI-2040 — GTI-2040 will be administered one day after HiDAC in the pilot PD study and one day before HiDAC in the Phase II study for a cycle. Those who achieve a complete remission (CR) will be permitted to receive one cycle of consolidation of GTI-2040 and HiDAC

SUMMARY:
This is a Phase II trial conducted at multiple centers for evaluation of the pharmacodynamic activity and the overall response rate contributed by the combination agents of GTI-2040 and High Dose Cytarabine (HiDAC) in Refractory and Relapsed Acute Myeloid Leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have unequivocal histologic diagnosis of AML according to WHO classification.
* Patients must have (1) refractory AML, defined as a disease unresponsive to the initial treatment; or (2) relapsed AML, defined as disease that re-occurs after treatment with conventional or high dose chemotherapy, with or without autologous stem cell support.
* Patients previously treated with antisense oligonucleotides remain eligible in absence of significant or dose-limiting documented toxicities directly attributable to the antisense agents.
* Age 18-59 years old.
* Because no dosing or adverse event data are currently available on the use of GTI-2040 in combination with cytarabine in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric Phase 2 combination trials.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2 (Karnofsky >60%).
* Patients with central nervous system (CNS) involvement will be considered eligible for this study if no residual leukemic cells are detectable in the cerebral spinal fluid following intrathecal or radiation therapy.
* Central line catheter for administration of GTI-2040 infusion is required for all patients enrolled in the study.
* Ability to understand and the willingness to sign a written informed consent document. Written informed consent is required prior to any study procedures for screening or enrollment.

Exclusion Criteria:

* Patients who have had chemotherapy (with the exception of hydroxyurea) or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Patients who have received mitomycin C or nitrosurea require a 6 week recovery period before enrollment.
* Patients who have had prior allogeneic stem cell transplant.
* Patients may not be receiving any other investigational agents as part of ongoing treatment.
* Patients with the following abnormal clinical values (unless abnormalities in these parameters are directly attributable to malignancy):

  * Resting cardiac ejection fraction < 50%
  * Serum creatinine > 1.5 mg/dL
  * Total bilirubin > 2x upper limits of normal (ULN) (unless due to Gilbert's syndrome)
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 3x ULN
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GTI-2040 or other agents used in the study.
* Patients who require chronic systemic anticoagulant therapy for medical conditions (e.g., previous history of deep venous thrombosis, atrial fibrillation etc.). Heparin administration to maintain central line patency (i.e. catheter flush) is not an exclusion.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Serious medical or psychiatric illness that would prevent informed consent or limit survival to < 4 weeks.
* Pregnancy or breastfeeding women. The potential for teratogenic effects and other risks for GTI-2040 in nursing infants are unknown. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
* HIV-positive patients on combination antiretroviral therapy are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca B Klisovic, MD, Principal Investigator — Ohio State University
Locations (7):
- United States (7):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Northside Hospital, Atlanta, Georgia
  - Indiana Cancer Research Institute, Indianapolis, Indiana
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Mount Sinai Hospital, New York, New York
  - The Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 acute myeloid leukemia (AML) patients with either relapse (> 6 months) after First complete remission (CR1) or refractory/early relapse CR1 duration < 6 months were enrolled into the study from 6 sites. In total, 25 patients were treated with GTI-2040.
Pre-assignment Details: Patients were enrolled in one of two treatment arms: "Pilot Arm" (Pilot PD Group) using delayed administration of GTI-2040, or a "Phase 2 Arm" (Phase II Group) using early administration of GTI-2040 with respect to High Dose Cytarabine (HiDAC).
Period: Overall Study
Arm/Group | Pilot | Phase II Arm
Started | 10 | 15
Completed | 9 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 27 acute myeloid leukemia patients with either relapse (> 6 months) after First complete remission (CR1) or refractory/early relapse CR1 duration < 6 months were enrolled into the study from 6 sites.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot | Phase II Arm | Total
Number analyzed (Participants) | 11 | 16 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 16 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 7 | 12 | 19
Region of Enrollment [Number; unit: participants]
  United States | 11 | 16 | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of GTI-2040 Combined With HiDAC in Refractory or Relapsed AML
Description: Overall Response was defined as whether or not the patient achieved complete remission (CR) and CR with incomplete blood count recovery (CRi) while on the study.
Time Frame: at 29-35 days
Population: All Treated Patients population
Measure: Number; unit: participants
Arm/Group | Pilot | Phase II Arm
Number analyzed (Participants) | 10 | 15
participants | 3 | 4

2. Secondary Outcome: Summary of Treatment Emergent Adverse Events
Description: An adverse event (AE) was defined as any unintended or undesirable experience that occurred during the course of the clinical investigation, regardless of whether or not it was considered to be study drug-related. This included any newly occurring event or a previous condition that had increased in severity or frequency since the administration of study drug.
Time Frame: 30 days after the last dose
Population: All Treated Patients population.
Measure: Number; unit: participants
Arm/Group | Pilot | Phase II Arm
Number analyzed (Participants) | 10 | 15
participants
  Number of Patients Reporting AEs | 10 | 15
  SAE | 2 | 2
  AE leading to Study Drug Discontinuation | 1 | 0
  Deaths within 30 days after the last dose of study | 1 | 0

ADVERSE EVENTS:
Time Frame: 310 days
Arm/Group | Pilot | Phase II Arm
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/15
Other Adverse Events (participants affected / at risk) | 10/10 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot (N=10) | Phase II Arm (N=15)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Disease Progression (General disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot (N=10) | Phase II Arm (N=15)
Anemia (Blood and lymphatic system disorders) | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 8
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 8
Lymphopenia (Blood and lymphatic system disorders) | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7
Tachycardia (Cardiac disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual disturbance (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 13
Oral mucosal petechiae (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 8
Asthenia (General disorders) | 0 | 1
Catheter site discharge (General disorders) | 1 | 0
Chills (General disorders) | 5 | 8
Disease progression (General disorders) | 2 | 0
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 7
Generalised oedema (General disorders) | 0 | 1
Infusion site erythema (General disorders) | 1 | 2
Infusion site haemorrhage (General disorders) | 0 | 1
Infusion site pain (General disorders) | 2 | 2
Mucosal inflammation (General disorders) | 3 | 2
Oedema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 7
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3
Bacteraemia (Infections and infestations) | 1 | 1
Candidiasis (Infections and infestations) | 1 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Central line infection (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Enterococcal infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Rash pustular (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 2
Streptococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 2
Blood albumin decreased (Investigations) | 3 | 0
Blood albumin increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood calcium decreased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 2 | 1
Blood uric acid increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 0 | 1
Clostridium difficile toxin test positive (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 1
International normalised ratio increased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 2 | 1
Protein total decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 2
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 3 | 9
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 3
Mood altered (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 3
Thrombophlebitis superficial (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less